CLINICAL TRIAL: NCT03644784
Title: Protocoled Quantitative Assessment of Aortic Regurgitation Using Videodensitometry in a Multicontinental Trial in Rotterdam, Montreal, Yamaguchi, Segeberg, Amsterdam.
Acronym: ASSESS-REGURGE
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Yamaguchi University Hospital (Other); Segeberger Kliniken GmbH (Other); McGill University (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Patrick W. Serruys, Prof. dr., Imperial College London
Other Study IDs: ASSESS-REGURGE
Record Dates: First submitted 2018-03-01; First posted 2018-08-23 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Aortic Valve Insufficiency; Aortic Valve Regurgitation
MeSH Terms: conditions — Aortic Valve Insufficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Yamaguchi University Hospital
  Interventions: Diagnostic Test: Standardized protocol for assessing aortic regurgitation using videodensitometry
- Erasmus Medical Center
  Interventions: Diagnostic Test: Standardized protocol for assessing aortic regurgitation using videodensitometry
- Academic Medical Center - Amsterdam
  Interventions: Diagnostic Test: Standardized protocol for assessing aortic regurgitation using videodensitometry
- Segeberger Kliniken Gruppe
  Interventions: Diagnostic Test: Standardized protocol for assessing aortic regurgitation using videodensitometry
- McGill University - Montreal
  Interventions: Diagnostic Test: Standardized protocol for assessing aortic regurgitation using videodensitometry

INTERVENTIONS:
Diagnostic Test: Standardized protocol for assessing aortic regurgitation using videodensitometry — Standardized protocol for assessing aortic regurgitation using videodensitometry

SUMMARY:
The ASSESS-REGURGE is a multicenter, multicontinental registry on protocoled aortographic image acquisition after implantation of a transcatheter aortic valve. After the implementation of the acquisition protocol, each participating site will use the standardized approach for their center in order to identify if the images are considered analyzable via videodensitometry quantitative assessment of aortic regurgitation.

ELIGIBILITY:
Inclusion Criteria:

* Eligible and undergoing TAVR procedure

Exclusion Criteria:

* Considered not eligible for TAVR procedure by the local Heart Team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with aortic regurgitation that are undergoing TAVR in the 5 centers
Sampling Method: Non-Probability Sample
Enrollment: 354 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Feasibility (percentage of the cases considered analyzable) of analysis of aortic regurgitation from aortograms using the videodensitometry technique | 1 year
  Measurement of feasibility, i.e. the percentage of the number of cases, out of the entire sample size that are considered to be analyzable for quantitative aortic regurgitation assessment using videodensitometry after the implementation of the acquisition protocol. Since the analyzability of the aortic regurgitation from the aortograms depends in some acquisition factors, we will assess the feasibility of analysis after implantation of acquisition protocols.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick W Serruys, MD, PhD, Study Chair — Imperial College London; Rodrigo Modolo, MD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Yoshinobu Onuma, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (6):
- McGill University, Montreal, Canada
- Segeberger Kliniken, Bad Segeberg, Germany
- Yamaguchi University, Yamaguchi, Japan
- Netherlands (2):
  - Academic Medical Center, Amsterdam
  - Erasmus Medical Center, Rotterdam
- Imperial College, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Modolo R, Chang CC, Tateishi H, Miyazaki Y, Pighi M, Abdelghani M, Roos MA, Wolff Q, Wykrzykowska JJ, de Winter RJ, Piazza N, Richardt G, Abdel-Wahab M, Soliman OII, Onuma Y, Van Mieghem NM, Serruys PW. Quantitative aortography for assessing aortic regurgitation after transcatheter aortic valve implantation: results of the multicentre ASSESS-REGURGE Registry. EuroIntervention. 2019 Aug 29;15(5):420-426. doi: 10.4244/EIJ-D-19-00362. PMID 31147307